CLINICAL TRIAL: NCT01024439
Title: Double Blinded Randomized Controlled Study of Conventional Laparoscopic Appendicectomy Versus Transumbilical Single Incision Laparoscopic Appendicectomy
Brief Title: Transumbilical Single Incision Versus Conventional Three Incisions Laparoscopic Appendicectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Kwok-Kay Yau, Specialist in general surgery, Pamela Youde Nethersole Eastern Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HKEC-2009-080
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- single port (Active Comparator): Patients will undergo transumbilical single incision laparoscopic appendicectomy.
  Interventions: Procedure: transumbilical single incision laparoscopic appendicectomy
- conventional Lap (Active Comparator): Patients will undergo conventional laparoscopic appendicectomy.
  Interventions: Procedure: conventional laparoscopic appendicectomy

INTERVENTIONS:
Procedure: transumbilical single incision laparoscopic appendicectomy — Patients will undergo transumbilical single incision laparoscopic appendicectomy. A single incision is made on umbilicus within the margin of umbilical skin ring. Peritoneal cavity is entered by open method and the fascia layer can be extended up to 2.5cm in length. A single incision laparoscopic device (Olympus) will be inserted. Conventional laparoscopic instruments will be used. Umbilical fascia will be closed by PDS-1 J-shape needle. Marcain 0.5% should be infiltrated into the fascial layers as well as the skin layers with dosage up to 20ml. The umbilicus is reconstructed by interrupted 3-0 nylon by tacking the skin onto the fascia layers.
  Three non-transparent dressings will be placed as if conventional laparoscopic appendicectomy has been done.
  Arms: single port
Procedure: conventional laparoscopic appendicectomy — Patients will undergo conventional laparoscopic appendicectomy. A 10-mm subumbilical port will be inserted by open method. Two 5-mm working ports will be inserted under laparoscopic view at patient's left lower quadrant and suprapubic area. Umbilical fascia will be closed by PDS-1 J-shape needle.
  Local anaesthetic agent , Marcain 0.5% should be infiltrated into the fascial layers as well as the skin layers with dosage up to 20ml. All skin wound will be approximated with 3-0 nylon interrupted stitches and covered with non-transparent dressings.
  Arms: conventional Lap

SUMMARY:
Laparoscopic appendicectomy is widely practiced in Hong Kong nowadays with shorter hospital stay and less wound complications. Most of the time, three small wounds of less than 10mm will be adequate enough for the completion of the surgery with minimal pain.

Recently, the concept of Natural Orifice Transluminal Endoscopic Surgery (N.O.T.E.S) led to the attention of single incision laparoscopic surgery (SILS) again in the surgical community. SILS is not a new idea. The first SILS for cholecystectomy was reported in 1997 by Navarra et al. However, the close proximity of the instruments, limitation in triangulation during dissection and suboptimal exposure of the surgical field has made this approach unpopular in last decade. Because the concept of N.O.T.E.S and the newly designed access port, surgeons are now focused again on SILS. The Chinese University of Hong Kong has recently release their preliminary results on the use of SILS on appendicectomy with satisfactory results in terms of less post-operative pain and less prominent scar. However, it was a case series with limited number of patients. In order to test the advantages of SILS on the management of patients with acute appendicitis, a double blinded randomized clinical trial is conducted.

DETAILED DESCRIPTION:
Double Blinded Randomized controlled study of Conventional Laparoscopic Appendectomy Vs Transumbilical Single Incision Laparoscopic Appendicectomy

Introduction:

Laparoscopic appendicectomy is widely practiced in HA hospital nowadays with shorter hospital stay and less wound complications. Most of the time, three small wounds of less than 10mm will be adequate enough for the completion of the surgery with minimal pain.

Recently, the concept of Natural Orifice Transluminal Endoscopic Surgery (N.O.T.E.S) led to the attention of single incision laparoscopic surgery (SILS) again in the surgical community[1,2,3] is not a new idea. The first SILS for cholecystectomy was reported in 1997 by Navarra et al. However, the close proximity of the instruments, limitation in triangulation during dissection and suboptimal exposure of the surgical field has made this approach unpopular in last decade. Because the concept of N.O.T.E.S and the newly designed access port, surgeons are now focused again on SILS. The Chinese University of Hong Kong has recently release their preliminary results on the use of SILS on appendicectomy with satisfactory results in terms of lesser post-operative pain and less prominent scar. However, it was a cases series with limited number of patients. In order to test the advantages of SILS on the management of patients with acute appendicitis, a double blinded randomized clinical trial is conducted.

Statistical Analysis:

The primary outcome that the trial to evaluate is operative time, post-operative pain and wound infection rate. The working alternative hypothesis is that there will be significant differences in umbilical wound infection rate between Conventional Laparoscopic Appendectomy and Transumbilical Single Incision Laparoscopic Appendicectomy.

At least 80 patients (40 cases in each group) is needed to demonstrate a 25% difference in umbilical wound infection rate at a statistical significance level of P> 0.05 and power of 80%. All analyses and comparisons between the two groups were performed on an intention-to-treat basis.

The Student t-test, Mann-Whitney U test, the Chi-square test and Fisher exact test where appropriate were used to compare the result between groups. All calculations were performed by the software SPSS for Window version 15.0 (SPSS, Inc, USA). P <0.05 was considered as statistical significant.

Detailed Description:

This study seeks to examine the ability of single incision laparoscopic appendicectomy to reduce the post-operative pain and increase cosmetic outcome at the expense of longer operation time and at higher cost. Patients will be randomized preoperatively by a computer generated random allocation to either receive conventional laparoscopic appendicectomy or to have transumbilical single incision laparoscopic appendicectomy.

Control group:

Patients will undergo conventional laparoscopic appendicectomy. A 10-mm subumbilical port will be inserted by open method. Two 5-mm working ports will be inserted under laparoscopic view at patient's left lower quadrant and suprapubic area. Umbilical fascia will be closed by PDS-1 J-shape needle.

Local anaesthetic agent , Marcain 0.5% should be infiltrated into the fascial layers as well as the skin layers with dosage up to 20ml. All skin wound will be approximated with 3-0 nylon interrupted stitches and covered with non-transparent dressings.

Compare group:

Patients will undergo transumbilical single incision laparoscopic appendicectomy. A single incision is made on umbilicus within the margin of umbilical skin ring. Peritoneal cavity is entered by open method and the fascia layer can be extended up to 2.5cm in length. A single incision laparoscopic device (Olympus) will be inserted. Conventional laparoscopic instruments will be used. Umbilical fascia will be closed by PDS-1 J-shape needle. Marcain 0.5% should be infiltrated into the fascial layers as well as the skin layers with dosage up to 20ml. The umbilicus is reconstructed by interrupted 3-0 nylon by tacking the skin onto the fascia layers.

Three non-transparent dressings will be placed as if conventional laparoscopic appendicectomy has been done.

Randomization:

Randomization is performed before consent for surgery. Patients are randomly assigned by means of sealed envelopes containing computer-generated random numbers into the following groups:

1. Control group (conventional laparoscopic appendicectomy)
2. Compare group (single port laparoscopic appendicectomy)

ELIGIBILITY:
Inclusion Criteria:

* Patients will be at least 18 years of age.
* Male or female (excluding pregnant females).
* Patients with ASA ≦ 3.
* Patients informed about the study, and will have read; understood and signed the patient informed consent. Patients will be willing and able to submit to postoperative follow-up evaluations.

Exclusion Criteria:

* Patients have previous history of abdominal surgery.
* Patients with ASA > 3.
* Patients with any conditions that were not suspected preoperatively and are only discovered at the time of the operation.
* Patients who are incompetent in giving consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
wound infection rate | 2 weeks after surgery

SECONDARY OUTCOMES:
cosmetic satisfaction | 2 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Pamela Youde Nethersole Eastern Hospital, Hong Kong, Hong Kong, China